CLINICAL TRIAL: NCT07073664
Title: A Prospective, Randomized, Single-blind, Self-controlled Study Evaluating the Efficacy of Endoscope Ethmoid Infundibulum Expansion Surgery (EEIES) Combined With Stapokibart in the Treatment of Type 2 Chronic Rhinosinusitis
Brief Title: A Study Evaluating the Efficacy of Endoscope Ethmoid Infundibulum Expansion Surgery (EEIES) Combined With Stapokibart in the Treatment of Type 2 Chronic Rhinosinusitis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Union Hospital (Other)
Responsible Party: Principal Investigator, Dongdong Zhu, Department Director, China-Japan Union Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2025041701
Record Dates: First submitted 2025-07-10; First posted 2025-07-18 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Chronic Sinusitis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The surgical side of Endoscope Ethmoid Infundibulum Expansion Surgery (EEIES) (Experimental)
  Interventions: Procedure: The surgical side of Endoscope Ethmoid Infundibulum Expansion Surgery (EEIES)
- The surgical side of Endoscopic Sinus Surgery (ESS) (Active Comparator)
  Interventions: Procedure: The surgical side of Endoscopic Sinus Surgery (ESS)

INTERVENTIONS:
Procedure: The surgical side of Endoscope Ethmoid Infundibulum Expansion Surgery (EEIES) — Surgery was performed by Endoscope Ethmoid Infundibulum Expansion Surgery (EEIES) . Stapokibart from two weeks after the operation, subcutaneous injection of Stapokibart was administered once every two weeks for six consecutive months, a total of 12 times.
  Arms: The surgical side of Endoscope Ethmoid Infundibulum Expansion Surgery (EEIES)
Procedure: The surgical side of Endoscopic Sinus Surgery (ESS) — Description: Surgery was performed by Endoscopic Sinus Surgery (ESS). Stapokibart from two weeks after the operation, subcutaneous injection of Stapokibart was administered once every two weeks for six consecutive months, a total of 12 times.
  Arms: The surgical side of Endoscopic Sinus Surgery (ESS)

SUMMARY:
Through a prospective study, the efficacy of Endoscope Ethmoid Infundibulum Expansion Surgery (EEIES) in the surgical treatment of patients with type 2 chronic rhinosinusitis was verified. The aim was to provide evidence-based medical evidence for the effectiveness of local minimally invasive surgery combined with biologics in the treatment of type 2 chronic rhinosinusitis.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnostic criteria for chronic rhinosinusitis refer to "Chinese Guidelines for Diagnosis and Treatment of Chronic Rhinosinusitis (2024)", namely: (1) Symptoms: nasal congestion, nasal discharge; secondary symptoms: headache in the head and face, reduced or lost sense of smell. (2) Endoscopic examination: bilateral lesions, mucous or mucopurulent secretions from the middle meatus and choana, nasal mucosa congestion, edema or polyps. The difference in endoscopic scores between both sides is no more than 2. (3) Imaging examination: bilateral lesions, nasal sinus CT scan can show the ostiomeatal complex and/or inflammatory lesions of the nasal sinus mucosa. The difference in CT scores between both sides is no more than 2.
2. Diagnostic criteria for type 2 chronic rhinosinusitis refer to "2023 EPOS on the indications for biological therapy of CRSwNP", namely: (1) Evidence of type 2 inflammation: eosinophils (EOS) >=10/hpf in tissue, or EOS>=150 in blood, or total IgE >=100; (2) Need for systemic glucocorticoids or contraindications to systemic glucocorticoids: >= 2 courses per year, or long-term (> 3 months) low-dose glucocorticoids; (3) Significant impairment of quality of life: SNOT-22 >= 40; (4) Obvious loss of sense of smell: loss of sense of smell in the smell test; (5) Diagnosis of combined asthma: asthma requiring regular inhalation of glucocorticoids. Three of the five conditions can diagnose type 2 inflammation.
3. History of rhinosinusitis for more than 2 years, patients enrolled in China-Japan Union Hospital of Jilin University whose residence is in Northeast China meet the requirements for postoperative follow-up (including Heilongjiang Province, Jilin Province, Liaoning Province, and Hulunbuir City, Xing'an League, Tongliao City, Chifeng City, and Xilingol League of Inner Mongolia Autonomous Region). Patients enrolled in the First Affiliated Hospital of Jinan University whose residence is in southern China meet the requirements for postoperative follow-up (including Guangdong Province and Guangxi Zhuang Autonomous Region).

Exclusion Criteria:

1. Pregnant women.
2. Patients with diabetes, hypertension, coronary heart disease, tuberculosis, asthma, and malignant tumors who cannot tolerate general anesthesia surgery.
3. Other patients who are unable to receive or unwilling to undergo surgical treatment due to severe systemic diseases or mental disorders.
4. Patients who are unable to cooperate with postoperative follow-up.
5. Age < 18 years old or > 75 years old.
6. Patients who have received allergen-specific immunotherapy or biological agent treatment within the past year.
7. Patients with a history of sinus surgery in the past.
8. Those with acute infectious diseases, upper respiratory tract infections or systemic inflammatory symptoms such as fever and chills.
9. Those who cannot tolerate severe systemic or local adverse reactions during relevant examinations or specimen collection.
10. Patients whom the researchers consider ineligible for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale(VAS) score of nasal symptoms | Two weeks, 1 month, 3 months, 6 months, and 12 months after surgery.
  The minimum possible scale value is 0, and the maximum possible scale value is 10. The higher scores mean a worse outcome.
Nasal endoscopy score(Lund-Kennedy scores, LKs) | Two weeks, 1 month, 3 months, 6 months, and 12 months after surgery.
  The minimum possible scale value is 0, and the maximum possible scale value is 10. The higher scores mean a worse outcome.
Paranasal sinus CT score(Lund-Mackey scores, LMs) | 6 months and 12 months after surgery.
  The minimum possible scale value is 0, and the maximum possible scale value is 12. The higher scores mean a worse outcome.
Nasal polyps scores(NPs) | Two weeks, 1 month, 3 months, 6 months, and 12 months after surgery.
  The minimum possible scale value is 0, and the maximum possible scale value is 4. The higher scores mean a worse outcome.
Questionnaire score for Sinusitis Quality of Life(SNOT-22 scores) | Two weeks, 1 month, 3 months, 6 months, and 12 months after surgery.
  The minimum possible scale value is 0, and the maximum possible scale value is 110. The higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Life quality score(SF-36 scores) | Two weeks, 1 month, 3 months, 6 months, and 12 months after surgery.
  The minimum possible scale value is 0, and the maximum possible scale value is 100. The higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Union Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Undecided